CLINICAL TRIAL: NCT06539988
Title: Advancing Decisions About Virtual Service Encounters (ADViSE)
Brief Title: Advancing Decisions About Virtual Service Encounters
Acronym: ADViSE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 22-172
Record Dates: First submitted 2024-06-26; First posted 2024-08-06 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Health Care Costs; Delivery of Health Care
Keywords: Access; Behavior (patient); Behavior (provider); Rural Health; Patient preferences; Decision support; Telemedicine; Patient-centered Care; Communication (doctor-patient); Cost; Patient outcomes; Primary care; Satisfaction (patient); Virtual care
MeSH Terms: conditions — Behavior; Patient Preference; Communication; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Receiving the optimized ADviSE Intervention (Experimental): 6 months of selected text messages from a library developed and refined in previous study aims.
  Interventions: Behavioral: Clinician Coaching Sessions; Other: Personalized text messages to patients
- Control period (No Intervention): Usual care.

INTERVENTIONS:
Behavioral: Clinician Coaching Sessions — PCPs will receive interactive coaching sessions from a Clinician Coach 2 months into the intervention period and again at 4 months into the intervention period.
  Arms: Receiving the optimized ADviSE Intervention
Other: Personalized text messages to patients — Drawing upon a library of messages that have previously been developed and refined, Veterans will receive 6 months of optimized text messages. The frequency of text messages will be determined based on feedback from Veterans in earlier phases of the research.
  Arms: Receiving the optimized ADviSE Intervention

SUMMARY:
Expanded availability of virtual care encounters in Primary Care provides new opportunities to improve Veterans' outcomes by aligning encounter modalities with their needs and preferences. Yet, Veterans and their Primary Care physicians (PCPs) lack personalized information about the benefits and costs of different Primary Care modalities that is needed to maximize the value of Primary Care encounters. To address this problem, in this study the investigators will use surveys and interviews to identify what Veterans and PCPs perceive to be the benefits and optimal uses of different Primary Care encounter modalities. They will then supplement their existing system for communicating encounter costs to Veterans and PCPs with new interactive messaging about benefits and optimal uses of different encounter modalities. Finally, this novel Advancing Decisions about Virtual Service Encounters (ADViSE) intervention will be optimized through user-centered refinement before evaluating its effects on Veteran-centered outcomes, use of virtual care, and intermediate health outcomes in a randomized controlled trial (RCT).

DETAILED DESCRIPTION:
The investigators will evaluate, in a stepped wedge cluster RCT, the effectiveness of the optimized ADViSE intervention, which will use interactive text messages for Veterans and point-of-care (POC) information and brief coaching for PCPs to help Veterans and their clinicians make well-informed decisions about available encounter types to meet each Veteran's needs and optimize the perceived value of their healthcare. A mixed methods stepped wedge cluster RCT will be conducted in which the optimized ADViSE intervention will be rolled out to PCPs and Veterans in each of 6 VA Ann Arbor Healthcare System (VAAAHS) Patient Aligned Care Teams (PACTs) in a randomly assigned order. For each Veteran participant, pre-post differences in outcomes during the 6-month intervention period will be compared to a 6-month pre-intervention control period.

ELIGIBILITY:
Inclusion Criteria:

* Veteran inclusion criteria are having an upcoming face-to-face (F2F), telephone, or VA Video Connect (VVC) appointment in the next 8 to 12 weeks
* Having at least 3 Primary Care F2F, telephone, or VVC encounters in the previous 12 months
* Able to provide informed consent
* Willing and able to receive text messages from the VA Patient Engagement, Tracking, and Long-term Support (PETALS) platform

Exclusion Criteria:

* Veteran exclusion criteria are a CDW diagnosis of mild cognitive impairment, dementia, or a psychotic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Veterans' perceptions of the value of their healthcare | 6 months prior to intervention and 6-months post intervention
  Measured by survey at baseline and intervention end

SECONDARY OUTCOMES:
VA Video Connect (VVC) encounters with assigned Patient Aligned Care Team (PACT) | 6 months prior to intervention and 6-months post intervention
  Measured using Corporate Data Warehouse (CDW) data
Face-to-Face (F2F) encounters with assigned Patient Aligned Care Team (PACT) | 6 months prior to intervention and 6-months post intervention
  Measured using CDW data
Telephone encounters with assigned Patient Aligned Care Team (PACT) | 6 months prior to intervention and 6-months post intervention
  Measured using CDW data
Veterans' satisfaction with healthcare | 6 months prior to intervention and 6-months post intervention
  Measured by survey at baseline and intervention end
Veterans' preferences for virtual care | 6 months prior to intervention and 6-months post intervention
  Measured by survey at baseline and intervention end
Total healthcare-associated costs for Veterans | 6 months prior to intervention and 6 months post intervention
  Sum of copay costs, travel costs, and time costs measured using CDW data
Hemoglobin A1c level <8% among Veterans with diabetes | 6 months prior to intervention and 6 months post intervention
  Electronic quality measure (eQM) measured using CDW data
Blood pressure (BP) < 140/90 among Veterans with diabetes | 6 months prior to intervention and 6 months post intervention
  Electronic quality measure (eQM) measured using CDW data
Statin use among Veterans with diabetes | 6 months prior to intervention and 6 months post intervention
  Electronic quality measure (eQM) measured using CDW data
Statin use among Veterans with ischemic heart disease | 6 months prior to intervention and 6 months post intervention
  Electronic quality measure (eQM) measured using CDW data
Breast cancer screening among female Veterans | 6 months prior to intervention and 6 months post intervention
  Electronic quality measure (eQM) measured using CDW data
Cervical cancer screening among female Veterans | 6 months prior to intervention and 6 months post intervention
  Electronic quality measure (eQM) measured using CDW data
Colon cancer screening among Veterans aged 45-75 | 6 months prior to intervention and 6 months post intervention
  Electronic quality measure (eQM) measured using CDW data
Flu vaccine receipt among Veterans | 6 months prior to intervention and 6 months post intervention
  Electronic quality measure (eQM) measured using CDW data
Time costs for Veterans | 6 months prior to intervention and 6 months post intervention
  Measured using CDW data
Travel costs for Veterans | 6 months prior to intervention and 6 months post intervention
  Measured using CDW data
Copay costs for Veterans | 6 months prior to intervention and 6 months post intervention
  Measured using CDW data

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey T. Kullgren, MD MPH MS, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No